CLINICAL TRIAL: NCT07232771
Title: Reinfection and Re-revision Rates of Periprosthetic Knee Infection Under Four Different Surgical Strategies: a Single Centre Retrospective Observational Study
Brief Title: Reinfection and Re-revision Rates of Periprosthetic Knee Infection Under Four Different Surgical Strategies
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Xinyu Fang, Deputy chief physician, First Affiliated Hospital of Fujian Medical University
Other Study IDs: MTCA,ECFAH of FMU[2019]296
Record Dates: First submitted 2025-09-27; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-09

CONDITIONS: Total Knee Arthroplasty; Reinfection; Aseptic Loosening; Revision; Periprosthetic Joint Infection (PJI)
Keywords: Total Knee Arthroplasty; Reinfection; Aseptic Loosening; Revision; Periprosthetic joint infection (PJI)
MeSH Terms: conditions — Reinfection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- DAIR group: DAIR revision involves washout, thorough debridement, antibiotics, and all components of implant retention, but polyethylene exchange
- 1-stage revision group: One-stage revision involves open debridement of the infected knee, followed by immediate revision by removal and or reimplantation of all components
- 1.5-stage revision group: The 1.5-stage revision involves the use of a functional, articulating antibiotic-loaded knee spacer intended for long-term retention-either indefinitely or until loosening necessitates definitive TKA revision. We standardize the terminology for this procedure as "1.5-stage revision", as it represents an intermediate strategy between one-stage and two-stage revision for the treatment of PJI following TKA
- 2-stage revision group: Two-stage revision, with removal of implants, placement of an antibiotic spacer, and parenteral antibiotic treatment followed by TKA reimplantation has been proposed as the "gold standard" for chronic PJI treatment

SUMMARY:
A single-center retrospective cohort study was conducted in the Department of Orthopedics, the First Affiliated Hospital of Fujian Medical University. This study reviewed 145 patients who underwent debridement, antibiotics, and implant retention (DAIR), 1-stage revision, 1.5-stage revision, and 2-stage revision surgeries for total knee arthroplasty periprosthetic joint infection (TKA-PJI) at this institution between 2012 and 2022. The differences in postoperative reinfection rate, microbial composition of reinfection, short-term and long-term aseptic prosthesis survival rate, prosthesis loosening and revision rate due to any cause, and long-term loosening-free survival rate among the four revision surgical approaches for TKA-PJI were evaluated, so as to provide reference value for clinical decision-making.

DETAILED DESCRIPTION:
A single-center retrospective cohort study was conducted in the Department of Orthopedics, the First Affiliated Hospital of Fujian Medical University. This study reviewed 145 patients who underwent debridement, antibiotics, and implant retention (DAIR), 1-stage revision, 1.5-stage revision, and 2-stage revision surgeries for total knee arthroplasty periprosthetic joint infection (TKA-PJI) at this institution between 2012 and 2022. In this study, we aimed to evaluate: (1) the postoperative reinfection rates following four surgical strategies for TKA-PJI; (2) the microbial profile of recurrent infections; (3) short- and long-term infection-free implant survival rates across the four surgical approaches; (4) re-revision rates due to aseptic loosening and long-term aseptic loosening-free implant survival rates; and (5) the reinfection rate in patients with positive cultures at the time of reimplantation. In order to provide reference value for clinical decision-making.

ELIGIBILITY:
Inclusion Criteria

1. Patients who met the diagnostic criteria for TKA-PJI;
2. Patients who underwent one of the following surgical interventions: DAIR, one-stage revision, 1.5-stage revision, or two-stage revision;
3. Patients with complete medical records available;
4. Patients who provided informed consent to participate in the study.

Exclusion Criteria:

1. Incomplete medical records;
2. Poor follow-up compliance, including inability to complete scheduled follow-up visits or refusal to participate in follow-up;
3. Follow-up duration less than 2 years.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: According to the inclusion criteria, 145 patients who underwent DAIR, phase 1 revision, phase 1.5 revision, and phase 2 revision surgery for TKA-PJI at the institution between 2012 and 2022 were selected. All patients have completed at least 2 years of follow-up. Follow up includes prosthesis loosening, infection recurrence rate, infection recurrence rate, infection new incidence rate, bacterial positive culture rate, infection free survival rate, and revision rate for any reason.
  Sampling Method
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Re-revision rate | 5 year after surgery
  Re-revisions with implant exchange
Reinfection rate | 2 and 5 year after surgery
  Reinfection rate
Infection-free survival rate | 2 and 5 year after surgery
  Infection-free survival rate
All-cause revision rates | 5 year after surgery
  All-cause revision rates

CONTACTS AND LOCATIONS:
Overall Officials: Liu Zhang, Study Director — First Affiliated Hospital of Fujian Medical University
Locations (1):
- The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China